CLINICAL TRIAL: NCT07374367
Title: Serum Isthmin-1 Level as a Biomarker of Disease Activity in Rheumatoid Arthritis: Correlation With Musculoskeletal Ultrasound Findings
Brief Title: Isthmin-1 as a Biomarker of Disease Activity in Rheumatoid Arthritis: Correlation With Musculoskeletal Ultrasound Findings
Status: Not yet recruiting | Type: Observational
Sponsor: Amera Imam Abdel - Ghany Ahmed (Other)
Responsible Party: Sponsor-Investigator, Amera Imam Abdel - Ghany Ahmed, Assistant lecturer, Assiut University
Organization: Assiut University (Other)
Other Study IDs: Isthmin-1, Rheumatoid ,MSUS
Record Dates: First submitted 2026-01-16; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Disease Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum sample of RA patients and controls to detect isthmin-1 level
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- rheumatoid arthritis patient
- age and sex matched healthy control

SUMMARY:
The goal of this case control study is to detect serum isthmin-1 level in RA patient compered to healthy control . The main questions it aims to answer are:

what is the serum isthmin-1 level in RA patient? what is the correlation between serum isthmin-1 and RA disease activity? what is the correlation between serum isthmin-1 level and MSUS finding in RA patients?

DETAILED DESCRIPTION:
Rheumatoid arthritis is a chronic autoimmune disease characterized by persistent synovitis, pannus formation, and bone erosion leading to joint damage and functional impairment . It manifests as a symmetrical polyarthritis predominantly affecting the small joints of the hands, the earliest and most severely affected site in RA. A total of 94% of the patients suffered from at least one hand or wrist symptom after 2-4 years of disease duration. The most frequently described symptoms were pain, stiffness of the hand, muscle weakness, paresthesia, and a limited fist, which significantly impair their daily hand function. Current monitoring tools, including ESR, CRP, and DAS-28, lack sensitivity for subclinical synovitis. These limitations underscore the need for novel biomarkers integrating systemic inflammatory activity with joint pathology and functional status.

Isthmin-1 (ISM1), a multifunctional adipokine that suppresses NF-κB pathway, thereby reducing pro-inflammatory cytokine production and promoting tissue repair . This mechanism holds relevance in RA, where aberrant NF-κB activation drives synovitis and Th17-mediated immune responses . Its observed reduction in active RA signifies a loss of endogenous anti-inflammatory counter-regulation, establishing ISM1 as a promising biomarker for disease activity monitoring .

Musculoskeletal ultrasound (MSUS) provides superior sensitivity compared to physical examination for detecting synovitis (. MSUS findings correlate with structural damage and functional decline, making it a valuable tool for monitoring disease impact on hand joints . This study investigates correlations between serum ISM1 levels, MSUS findings, and hand function to identify biological links for novel RA therapies that preserve joint function and enhance quality of life.

ELIGIBILITY:
Inclusion Criteria:

-Adult patients (≥18 years old) clinically diagnosed with rheumatoid arthritis according to the 2010 ACR/EULAR classification criteria.

Exclusion Criteria:

* Patients less than 18 years old.
* Patients with other autoimmune diseases.
* Participants with active infections, malignancies or diabetes.
* Recent hand surgery, trauma, deformity and neurological conditions affecting hand function

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years old) clinically diagnosed with rheumatoid arthritis according to the 2010 ACR/EULAR classification criteria.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Detection of serum isthmin-1 level in RA patients compared to healthy controls. | baseline
  The quantitative level of Human ISM1 will be measured with a commercial enzyme-linked immunosorbent assay(ELISA) kit.

SECONDARY OUTCOMES:
To correlate serum ISM1 levels with disease activity in RA | baseline
  through clinical and acute phase reactant

IPD SHARING:
Plan to Share IPD: No